CLINICAL TRIAL: NCT00003792
Title: Dendritic Cell Immunotherapy of Metastatic Melanoma - A Phase I Trial
Brief Title: Vaccine Therapy in Treating Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor Health Care System (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: BAYUMC-098004; CDR0000066935 (Registry Identifier: PDQ (Physician Data Query)); NCI-T98-0054
Record Dates: First submitted 1999-11-01; First posted 2004-07-16 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2006-10

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — MART-1 Antigen; Filgrastim; MAGEA3 protein, human

INTERVENTIONS:
Biological: MART-1 antigen
Biological: filgrastim
Biological: flu matrix peptide p58-66
Biological: gp100 antigen
Biological: recombinant MAGE-3.1 antigen
Biological: tyrosinase peptide
Procedure: in vitro-treated peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Vaccines made from a person's white blood cells and melanoma cells may make the body build an immune response and kill tumor cells.

PURPOSE: Phase I trial to study the effectiveness of vaccine therapy in treating patients who have metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety and tolerability of antigen pulsed dendritic cell therapy in patients with metastatic melanoma. II. Perform serial analysis of T cell and B cell function in these patients after this treatment. III. Determine objective response and response duration in these patients after this treatment.

OUTLINE: Patients receive filgrastim (G-CSF) subcutaneously (SQ) on days 1-6, then undergo leukapheresis for 2-3 days, beginning on day 6. Mononuclear cells are selected for CD34+ cells in the laboratory, made into dendritic cells, and then pulsed with MART-1, gp100, tyrosinase, MAGE-3 peptides and flu matrix. These antigen pulsed dendritic cells (ApDCs) are used for vaccinations. Prior to vaccination, ApDCs are mixed with MART-1, gp100, tyrosinase, MAGE-3, and flu matrix. Patients receive this dendritic cell vaccine mixture SQ every 2 weeks for 4 priming doses. Patients receive 4 boost vaccinations SQ at 2 months, 5 months, 9 months, and 15 months following the last priming vaccination. Patients are followed monthly for 2 years.

PROJECTED ACCRUAL: A total of 28 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven metastatic melanoma Measurable disease HLA-A2 01 phenotype No active CNS or hepatic metastases

PATIENT CHARACTERISTICS: Age: 18 to 80 Performance status: Karnofsky 80-100% Life expectancy: Not specified Hematopoietic: Normal CD4 and CD8 T cell numbers by flow cytometry Lactic dehydrogenase less than 2 times normal Hepatic: No viral hepatitis Renal: Not specified Cardiovascular: No prior venous thrombosis, angina pectoris, or congestive heart failure Pulmonary: No prior asthma Immunologic: Positive intradermal skin test for mumps, histoplasmosis, or streptokinase antigen Immunoglobulin levels normal No prior autoimmune disease (lupus erythematosus, rheumatoid arthritis, or thyroiditis) No allergy to tetanus toxoid or influenza vaccine No sensitivity to E. coli drug preparations Other: Not pregnant or nursing Fertile patients must use effective contraception HIV negative No active infection

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior interferon At least 8 weeks since prior interleukin-2 Chemotherapy: No more than 3 prior courses of cytotoxic chemotherapy At least 8 weeks since prior chemotherapy Endocrine therapy: No concurrent corticosteroids Radiotherapy: Not specified Surgery: Not specified Other: No other concurrent immunosuppressive agents

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-04; Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph W. Fay, MD, Study Chair — Baylor Health Care System
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States